CLINICAL TRIAL: NCT02683278
Title: Fibromyalgia: Interventions for Pain and Mood Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Mary Davis, Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AR053245 (NIH)
Record Dates: First submitted 2016-02-07; First posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive-Behavioral Therapy (Experimental): Group-based cognitive-behavioral manualized treatment
  Interventions: Behavioral: Cognitive-behavioral
- Mindfulness-acceptance Therapy (Experimental): Group-based mindfulness-acceptance manualized treatment
  Interventions: Behavioral: Mindfulness-acceptance
- Education (Active Comparator): Group-based manualized pain education
  Interventions: Other: Pain Education

INTERVENTIONS:
Behavioral: Cognitive-behavioral — Seven sessions of group-based treatment targeting skills to improve dysfunctional pain-related thoughts and behaviors
  Arms: Cognitive-Behavioral Therapy
Behavioral: Mindfulness-acceptance — Seven sessions of group-based treatment targeting skills to improve mindful awareness and acceptance of pain and stress, and increase positive emotional experiences
  Arms: Mindfulness-acceptance Therapy
Other: Pain Education — Seven sessions of group-based education to provide information regarding managing a chronic pain condition, but with no exercises to promote skill development
  Arms: Education

SUMMARY:
This study compares the impact of cognitive-behavioral therapy for pain (CBT-P), mindful awareness and acceptance treatment (M), and arthritis education as an active control condition (E) on mental and physical health outcomes among adults with chronic pain due to fibromyalgia (FM).

DETAILED DESCRIPTION:
Both cognitive-behavioral and mindful-acceptance based treatments impact pain and disability in people with chronic pain conditions like fibromyalgia. However, these treatments target different mechanisms. The focus of CBT is on helping individuals manage their thoughts and behaviors related to pain. In contrast, the focus of M is on improving individuals' ability be aware of and accept their experiences, and to develop their positive emotional resources.

ELIGIBILITY:
Inclusion Criteria:

* Pain in at least 11 of 18 tenderpoints
* Able to participate in study assessments and group-based meetings
* Willing to be randomized to treatment condition

Exclusion Criteria:

* Unable to understand written and spoken English
* Involved in pain-related litigation
* Currently involved in psychological treatment for pain and/or mood symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2008-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Physical Functioning | Change from baseline, 6-mo followup, and 12-mo followup
  Assessed via the SF-36 physical functioning subscale (Reference: Ware JE, Sherbourne CD. The MOS 36-Item Short-Form Health Survey (SF-36: I. conceptual framework and item selection. Med Care 1992; 30(6):473-83.
Bodily Pain | Change from baseline, 6-mo followup, and 12-mo followup
  Assessed via the SF-36 Bodily Pain subscale (Reference: Ware JE, Sherbourne CD. The MOS 36-Item Short-Form Health Survey (SF-36): I. conceptual framework and item selection. Med Care 1992; 30(6):473-83.
Vitality | Change from baseline, 6-mo followup, and 12-mo followup
  Assessed via the SF-36 Vitality subscale (Reference: Ware JE, Sherbourne CD. The MOS 36-Item Short-Form Health Survey (SF-36): I. conceptual framework and item selection. Med Care 1992; 30(6):473-83.
Depressive symptoms | Change from baseline, 6-mo followup, 12-mo followup
  Assessed via the Hamilton Depression Inventory (Reference: Reynolds WM, Kobak KA. Reliability and validity of the Hamilton Depression Inventory: A paper-and-pencil version of the Hamilton Depression Rating Scale Clinical Interview. Psychological Assessment 1995; 7(4): 472-83.
Social Functioning | Change from baseline, 6-mo followup, and 12-mo followup
  Assessed via the SF-36 Social Functioning subscale (Reference: Ware JE, Sherbourne CD. The MOS 36-Item Short-Form Health Survey (SF-36): I. conceptual framework and item selection. Med Care 1992; 30(6):473-83.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Davis, Ph.D., Principal Investigator — Arizona State University

IPD SHARING:
Plan to Share IPD: No